CLINICAL TRIAL: NCT03292939
Title: The Effect of Vaginal Progestrone on Fetal and Maternal Doppler Indices
Brief Title: Progestrone and Doppler Indices
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, sarah mohamed hassan, lecturer of obstetrics and gynecology Cairo university, Kasr El Aini Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 7880
Record Dates: First submitted 2017-09-20; First posted 2017-09-26 (Actual); Last update posted 2017-10-11 (Actual); Status verified 2017-10

CONDITIONS: Preterm Labor
Keywords: progestrone; doppler indices
MeSH Terms: conditions — Obstetric Labor, Premature

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- vaginal progestrone group (Other): cohort of patients who received 400mg vaginal progestrone .
  Interventions: Diagnostic Test: A complete Doppler ﬂow assessment of the maternal and fetal circulation

INTERVENTIONS:
Diagnostic Test: A complete Doppler ﬂow assessment of the maternal and fetal circulation — A complete Doppler ﬂow assessment of the maternal and fetal circulation was conducted by an independent investigator blinded to the treatment, 48 hours after receiving 400mg of vaginal progestrone .Voluson E8 (GE Healthcare, Zipf, Austria) ultrasound machine ,equipped with a 3.5-MHz curvilinear abdominal transducer with color imaging capabilities, was used in all cases.

SUMMARY:
The aim of our study is to assess the effect of vaginal progestrone on fetal and maternal doppler indices

DETAILED DESCRIPTION:
A complete Doppler ﬂow assessment of the maternal and fetal circulation was conducted by an independent investigator blinded to the treatment, before and 48 hours after the ﬁrst administration of 400mg of vaginal progesterone, Voluson E8 (GE Healthcare, Zipf, Austria) ultrasound machine,equipped with a 3.5- MHz curvilinear abdominal transducer with color imaging capabilities, was used in all cases.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age: 18-33 weeks
* Willing and able to give informed consent
* History of preterm labor (<34 weeks)
* At risk for preterm labor ( increased amniotic fluid volume)
* Short cervical length (<25mm) as incidental finding
* Presenting with actual cervical changes ( dilatation and\or effacement) in current pregnancy

Exclusion Criteria:

* PPROM
* Contraindication to progesterone use
* Diabetic patients, have glucose intolerance
* Multiple pregnancies

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-10-01 (Actual); Study Completion 2017-10-01 (Actual)

PRIMARY OUTCOMES:
change of ultrasound doppler indices. | before and 48 hours after progestrone admistration
  A complete Doppler ﬂow assessment of the maternaland fetal circulation was conducted by an independent investigator blinded to the treatment, before and 48 hours after the ﬁrst administration of progesterone, Voluson E8 (GE Healthcare, Zipf, Austria) ultrasoundmachine,equippedwitha3.5-MHzcurvilinearabdominaltransducer with color imaging capabilities, was used in all cases.

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr El Ainiy Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No